CLINICAL TRIAL: NCT06298695
Title: Cost-effectiveness of Schema Therapy for Treatment-resistant Anxiety Disorders: A Multicentre RCT
Brief Title: Schema Therapy for Treatment-resistant Anxiety Disorders
Acronym: PaDoLA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); ADF Stichting (Unknown); University of Amsterdam (Other); Maastricht University (Other); GGZ inGeest (Other); Pro Persona Mental Health Care Foundation (Other); Mondriaan (Unknown); GGNet (Unknown); GGZ Delfland (Unknown)
Responsible Party: Principal Investigator, Anna Muntingh, PhD, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012939; 10390022210010 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2024-02-29; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Anxiety Disorders
Keywords: agoraphobia; social anxiety disorder; generalized anxiety disorder; panic disorder; specific phobia; separation anxiety disorder; treatment-resistance; schema therapy; randomized controlled trial; cost-effectiveness
MeSH Terms: conditions — Anxiety Disorders; Agoraphobia; Phobia, Social; Generalized Anxiety Disorder; Panic Disorder; Phobia, Specific; Anxiety, Separation

STUDY DESIGN:
Intervention Model Description: A multicenter parallel group randomized controlled clinical intervention trial
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual Schema Therapy (Experimental): A maximum of 40 sessions of individual schema therapy within one year
  Interventions: Behavioral: Individual Schema Therapy
- Treatment As Usual (TAU) (Active Comparator): Treatment as usual in treatment-resistant anxiety disorders (psychological and/or psychiatric).
  Interventions: Other: TAU

INTERVENTIONS:
Behavioral: Individual Schema Therapy — Schema therapy focuses on adapting maladaptive "schemas" (i.e., core representations of oneself, others or the world) and dysfunctional personality traits, while also incorporating exposure therapy. It consists of a maximum of 40 sessions within one year.
  Arms: Individual Schema Therapy
Other: TAU — Treatment As Usual according to the Dutch Multidisciplinary Guidelines Anxiety Disorders and the Dutch Quality Standard for Anxiety Disorders. TAU often consists of a continuation of Cognitive Behavioral Therapy (CBT) and (different) medications, sometimes in a more treatment-intensive format. There are no restrictions to TAU, except that it may not be schema therapy. The actual content of TAU will be tracked.
  Arms: Treatment As Usual (TAU)

SUMMARY:
The aim of this study is to assess the cost-effectiveness of schema therapy compared to treatment as usual (TAU) in patients with treatment-resistant anxiety disorders. In a multicenter randomized controlled trial, patients will be assigned to receive individual schema therapy (maximum of 40 sessions) or treatment as usual (control group) within one year. The primary outcome is the difference between ST and TAU conditions in anxiety symptoms as measured with the Beck Anxiety Inventroy (BAI) at post treatment. Secondary outcomes include quality of life, societal costs, general mental health, remission from the anxiety disorders and/or comorbid affective disorders, positive and negative effects of psychotherapy, schemas and schema modes, and satisfaction. Measurements take place at baseline and after 1, 3, 6, 12, 24 and 36 months (follow-up of two years).

DETAILED DESCRIPTION:
RATIONALE Although treatment for anxiety disorders is generally (cost-)effective, a significant proportion of 30 to 60% of patients does not adequately respond to first-line treatments (i.e. cognitive behavioral therapy (CBT) and antidepressants). This patient group remains significantly impaired. A next-step psychotherapy focusing on underlying vulnerability is urgently needed.

OBJECTIVE To evaluate the cost-effectiveness of individual schema therapy (max. 40 sessions) versus treatment as usual in patients with treatment-resistant anxiety disorders from a societal perspective.

STUDY DESIGN Multicenter randomized controlled trial with a cost-effectiveness analysis and an embedded process evaluation. The project title "PaDoLA" refers to "PAtronen DOorbreken bij Langdurige Angst" in Dutch, which translates to "breaking patterns in chronic anxiety".

STUDY POPULATION Adults (18-65 years) with treatment-resistant DSM-5 anxiety disorders recruited in specialized mental health care. Treatment-resistance is defined as (at least) one failed trial of > 8 weeks CBT plus one failed trial of a serotonergic antidepressant for > 8 weeks plus persistence of anxiety symptoms.

INTERVENTION Intervention group: Individual schema therapy with max. 40 sessions within one year. Schema therapy is an integrative psychotherapy, with a high emphasis on the therapeutic relationship ("limited reparenting"), use of trauma focused techniques, experiential and cognitive techniques, role-play and behavioral exercises. The treatment protocol used in this study is adapted specifically for patients with treatment-resistant anxiety disorders.

Control group: Treatment as usual (TAU) described by the Dutch Quality Standard for Anxiety disorders. As there is no gold standard psychotherapy for treatment-resistant anxiety disorders, professionals often offer (extended or intensified) CBT and/or pharmacological treatment in TAU. The only restriction to TAU is that schema therapy may not be provided.

MAIN STUDY PARAMETERS/ENDPOINTS:

Primary outcome is the difference in anxiety symptoms as measured with the BAI at post treatment. Primary outcomes for the cost-effectiveness analysis are anxiety symptoms, quality of life and (societal) costs. Measurements take place at baseline and after 1, 3, 6, 12, 24 and 36 months. Secondary outcomes are general mental health, remission from the anxiety disorders and/or comorbid affective disorders, positive and negative effects of psychotherapy, schemas and schema modes, and satisfaction. Alongside the RCT, a process evaluation is performed to gain insight in experiences of patients and provide suggestions for implementation.

SAMPLE SIZE/DATA ANALYSIS A total of 172 patients will be enrolled (assuming a medium effect size d=0.5, testing two-sided using at ɑ=0.05, power = 0.80) including adjustment for an anticipated 25% dropout. We will perform an intention-to-treat analysis using a linear mixed model.

COST-EFFECTIVENESS ANALYSIS A cost-effectiveness and cost-utility analysis will be performed to compare effects on anxiety symptoms, quality of life and costs from a societal perspective including health care costs and productivity costs.

TIME SCHEDULE Study duration is 7 years: the first four years preparations will be made, patients will be included and treated. The follow-up phase of 2 years is necessary because effects are expected to be most prominent in the long term. Implementation efforts will be continuous during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of an anxiety disorder (panic disorder, agoraphobia, social anxiety disorder, generalized anxiety disorder, separation anxiety disorder and specific phobia) based on the Diagnostic and Statistical Manual of Mental Disorders (DSM-5).
* Fulfilling the criteria of treatment-resistance based on a systematic literature search by Bokma and collegues: i) at least one unsuccessful CBT treatment of ≥ 8 weeks; and ii) at least one unsuccessful pharmacological treatment with a serotonergic antidepressant of ≥ 8 weeks, and iii) moderate to severe anxiety symptoms (BAI > 11). The adequacy of previous treatment will be checked.

Exclusion Criteria:

* Substance use dependence
* Acute suicidality
* Has received schema therapy in the past
* Has insufficient language skills in Dutch and/or English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the severity of anxiety symptoms | Screening, baseline and at 1, 3, 6, 12, 24 and 36 months after baseline.
  Changes in the severity of anxiety symptoms are measured with the 21-item self-report Beck Anxiety Inventory (BAI), assessing somatic and affective-cognitive symptom domains. The total score ranges from 0 to 63, with higher scores indicating more severe anxiety symptoms. A score above 11 indicates clinically significant symptoms.
Health-related quality of life | Baseline and at 1, 3, 6, 12, 24 and 36 months after baseline.
  Health-related quality of life, which is used for the cost-utility analysis, is assessed with the 5-item, self-report Health-Related Quality of Life Measure Euroqol (EQ5D-5L). The EQ5D-5L measures five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The dimension scores can be translated into a single index value. Additionally, the EQ5D-5L estimates the general self-reported health-related quality of life on a visual analogue scale, ranging from 0 (worst quality of life) to 100 (best quality of life).
Mental health quality of life | Baseline and at 1, 3, 6, 12, 24 and 36 months after baseline.
  Mental health quality of life, which is used for the cost-utility analysis, is measured with the 7-item, self-report Mental Health Quality of Life (MHQoL). The MHQoL encompasses seven dimensions: self-image, independence, mood, relationships, daily activities, physical health and hope. Total scores range from 0 to 21, with higher scores indicating better quality of life. In addition, the MHQoL assesses self-reported general psychological well-being on a visual analogue scale, ranging from 0 (low well-being) to 10 (high well-being).
Health care utilization and productivity losses | Baseline and at 1, 3, 6, 12, 24 and 36 months after baseline.
  Health care utilization and productivity losses, which are used for the cost-utility analysis, are assessed with the 57-item, self-report Treatment Inventory of Costs in Patients with psychiatric disorders (TiC-P). The TiC-P measures two dimensions: health care use in psychiatric patients and (voluntary) work and care tasks. The IMTA Productivity Cost Questionnaire (iPCQ) is part of the TiC-P questionnaire and measures absenteeism, presenteeism and productivity loss in unpaid work.

SECONDARY OUTCOMES:
Remission from the primary anxiety disorder and from comorbid disorders | Baseline, and at 12, 24 and 36 months after baseline.
  Remission from the primary anxiety disorder and from comorbid disorders are measured with the short diagnostic Mini-International Neuropsychiatric Interview (MINI-S), which assesses mood disorders, anxiety disorders, OCD, PTSD, substance abuse, suicidal thoughts/behaviors and psychotic disorders. The interview is used for screening, assessing all of these disorders to check inclusion and exclusion criteria. It is also used in follow up to assess remission of the anxiety disorder and related disorders (anxiety, mood, OCD and PTSD).
Screening for DSM-5 personality disorders | Baseline and at 1, 3, 6, 12, 24 and 36 months after baseline.
  The 106-item, self-report Structured Clinical Interview DSM-5 Screening Personality Questionnaire (SCID-5-SPQ) is used for screening for DSM-5 personality disorders. The SCID-5-SPQ assesses the following personality disorders: paranoid, schizoid, schizotypal, antisocial, borderline, histrionic, narcissistic, avoidant, dependent and obsessive-compulsive personality disorder. Based on the SCID-5-SOQ the relevant personality disorders are assessed with the SCID-5-PD interview.
Assessment of DSM-5 personality disorders | Baseline
  The diagnostic interview SCID-5-PD is administered to assess DSM-5 personality disorders. The SCID-5-PD assesses the following personality disorders: paranoid, schizoid, schizotypal, antisocial, borderline, histrionic, narcissistic, avoidant, dependent and obsessive-compulsive personality disorder.
Demographics | Baseline
  Various demographics are collected: gender, age, ethnic background, socio-economic status, living situation, sexual orientation and educational level.
(Strength of) treatment preference | Baseline and at 12 months after baseline.
  Participants will be asked to rate their preference for schema therapy or TAU on a visual analogue scale ranging from a very strong preference for TAU to a very strong preference for schema therapy.
Assessment of childhood trauma | Baseline
  Childhood trauma is assessed with the 10-item, self-report Adverse Childhood Experiences (ACE) questionnaire. The ACE measures ten types of adverse childhood experiences, including negative experiences relating to themselves (i.e., physical, sexual and verbal abuse, and psychical and emotional neglect) and negative experiences relating to their family (i.e., domestic violence among parents/adults, alcoholic parents/adults, family members in prison, family members with a mental disorder, and the disappearance of a parent because of divorce, death or abandonment). The total score ranges from 0 to 10, with higher scores indicating more childhood trauma. A score above 4 indicates a clinically significant score.
Assessment of autistic traits | Baseline
  Autistic traits are measured with the 10-item, self-report Autism Spectrum Quotient short version (AQ-10). The total score ranges from 0 to 10. A score above 6 is considered clinically significant
Assessment of general mental health | Baseline and at 12, 24 and 36 months after baseline.
  General mental health is assessed with the 48-item, self-report Symptom Questionnaire-48 (SQ-48). The SQ-48 consists of nine different subscales: Depression, Anxiety, Somatisation, Agoraphobia, Aggression, Cognitive problems, Social Phobia, Work functioning, and Vitality. The SQ-48 includes items on suicidal thoughts. The total score ranges from 0 to 148 (without the subscales "work functioning" and "vitality"), with higher scores indicating poorer general mental health.
Functioning and recovery in psychiatric patients | Baseline and 12, 24 and 36 months after baseline.
  Functioning and recovery in psychiatric patients are measured with the 12-item, self-report individual Recovery Outcomes Counter (iROC). The iROC consists of four dimensions: home, people, opportunity, and empowerment. Higher (mean) scores indicate higher well-being.
Early Maladaptive Schemas | Baseline and at 12 and 36 months after baseline.
  Early Maldaptive Schemas (EMS) are assessed with the 90-item, self-report Young Schema Questionnaire 3 Short Form (YSQ-S3). The YSQ-3 measures all eighteen schemas. Total scores range from 90 to 540. Additionally, the mean score for each schema is calculated.
Schema Modes | Baseline and at 3, 6, 12 and 36 months after baseline.
  Schema Modes are measured with the 174-item, self-report Schema Mode Inventory 2 (SMI-2). The SMI assesses the strength of 18 adaptive and maladaptive schema modes.
Positive and negative effects of psychotherapy | At 12 months after baseline.
  The positive and negative effects of psychotherapy are measured with the 73-item, self-report Positive and Negative Effects of Psychotherapy questionnaire (PNEP). The PNEP contains 36 items regarding negative effects and 33 items regarding positive effects of psychotherapy.
The level of satisfaction with the psychological treatment | At 12 months after baseline.
  The level of satisfaction with the psychological treatment is measured with the 8-item, self-report Client Satisfaction Questionnaire (CSQ-8). The total score ranges from 8 to 32, with higher scores indicating more satisfaction with the treatment.

IPD SHARING:
Plan to Share IPD: No